CLINICAL TRIAL: NCT05549401
Title: A Phase I Clinical Trial to Evaluate the Tolerability and the Pharmacokinetics of CKD-348 With Co-administration of CKD-828, D097, and D337 in Healthy Adult Volunteers
Brief Title: Clinical Trial to Evaluate the Tolerability and the Pharmacokinetics of CKD-348
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A86_11BE2218P
Record Dates: First submitted 2022-09-18; First posted 2022-09-22 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Hypertension and Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Period 1: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition Period 2: CKD-348(4) F1 - A single oral dose of 1 tablet under fasting condition Period 3: CKD-348(4) F2 - A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-348(4) F1; Drug: CKD-348(4) F2; Drug: CKD-828, D097, D337
- Sequence 2 (Experimental): Period 1: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition Period 2: CKD-348(4) F2 - A single oral dose of 1 tablet under fasting condition Period 3: CKD-348(4) F1 - A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-348(4) F1; Drug: CKD-348(4) F2; Drug: CKD-828, D097, D337
- Sequence 3 (Experimental): Period 1: CKD-348(4) F1 - A single oral dose of 1 tablet under fasting condition Period 2: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition Period 3: CKD-348(4) F2 - A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-348(4) F1; Drug: CKD-348(4) F2; Drug: CKD-828, D097, D337
- Sequence 4 (Experimental): Period 1: CKD-348(4) F1 - A single oral dose of 1 tablet under fasting condition Period 2: CKD-348(4) F2 - A single oral dose of 1 tablet under fasting condition Period 3: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition
  Interventions: Drug: CKD-348(4) F1; Drug: CKD-348(4) F2; Drug: CKD-828, D097, D337
- Sequence 5 (Experimental): Period 1: CKD-348(4) F2 - A single oral dose of 1 tablet under fasting condition Period 2: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition Period 3: CKD-348(4) F1 - A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-348(4) F1; Drug: CKD-348(4) F2; Drug: CKD-828, D097, D337
- Sequence 6 (Experimental): Period 1: CKD-348(4) F2 - A single oral dose of 1 tablet under fasting condition Period 2: CKD-348(4) F1 - A single oral dose of 1 tablet under fasting condition Period 3: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition
  Interventions: Drug: CKD-348(4) F1; Drug: CKD-348(4) F2; Drug: CKD-828, D097, D337

INTERVENTIONS:
Drug: CKD-348(4) F1 — QD, PQ
Drug: CKD-348(4) F2 — QD, PQ
Drug: CKD-828, D097, D337 — QD, PQ

SUMMARY:
A phase I clinical trial to evaluate the tolerability and the pharmacokinetics of CKD-348.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged ≥ 19 years
2. Weight ≥55kg with calculated body mass index (BMI) of 18 to 30 kg/m2
3. Those who meet the blood pressure criteria during screening tests:

   * Systolic Blood Pressure: 90 to 139 mmHg
   * Diastolic Blood Pressure: 60 to 89 mmHg
4. Those who have no congenital diseases or chronic diseases and have no abnormal symptoms or findings.
5. Those who are eligible for clinical trials based on laboratory (hematology, blood chemistry, serology, urology) and 1ECG results at screening.
6. Those who agree to contraception during the participation of clinical trial.
7. Individuals who voluntarily decide to participate and agree to comply with the cautions after fully understand the detailed description of this clinical trial.

Exclusion Criteria:

1. Those who received investigational products or participated in bioequivalence tests within 6 months before the first administration of clinical trial drugs.
2. Those who take barbiturate and any related drugs which may cause induction or inhibition of drug metabolism within 1 month and those who take drug could affect to clinical trial within 10 days before the first administration of investigational products.
3. Those who donated whole blood or apheresis within 8 weeks or 4 weeks respectfully, or received blood transfusion within a month.
4. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery.
5. Those who exceed an alcohol and cigarette consumption criteria write below within 1 month before the first administration of investigational products.

   * Alcohol: Man - 21 glasses/week Woman - 14 glasses/week (1 glass: Soju 50mL, Wine 30mL, or beer 250mL)
   * Smoking: 20 cigarettes/day
6. Those who have any history of diabetic mellitus, nephropathy, biliary obstruction, shock, angioedema, cardiac insufficiency, dihydropyridine sensitivity, unstable angina, hypothyroidism.
7. Those who have genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption.
8. Those who are deemed insufficient to participate in this clinical trial by investigators.
9. Woman who are pregnant or breastfeeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-348(4) F1 and CKD-348(4) F2 | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  AUCt: Area under the concentration-time curve from time zero to time
Cmax of CKD-348(4) F1 and CKD-348(4) F2 | Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours
  Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Jaewoo Kim, M.D. Ph.D, Principal Investigator — m3116@newyjh.com
Locations (1):
- H plus Yangji hospital, Seoul, South Korea